CLINICAL TRIAL: NCT00827879
Title: Strength at Home Couples Program (Formerly: PTSD-Focused Relationship Enhancement Therapy for Returning Veterans and Their Partners)
Brief Title: Strength at Home Couples Program (PTSD-Focused Relationship Enhancement Therapy for Returning Veterans)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston VA Research Institute, Inc. (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Casey Taft, Principal Investigator, Boston VA Research Institute, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: U49CE001248 (NIH)
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Aggression; Post Traumatic Stress Disorders
Keywords: Intimate partner aggression; Couples intervention; PTSD; Veterans; Prevention; Violence Prevention; Prevention of pertetration of intimate partner aggression.
MeSH Terms: conditions — Aggression; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Strength at Home Couples Group (Experimental): PTSD-Focused Cognitive Behavioral Therapy for Couples
  Interventions: Behavioral: Strength at Home Couples Group
- Supportive Group Therapy (Placebo Comparator): Supportive therapy for couples
  Interventions: Behavioral: Supportive Group Therapy

INTERVENTIONS:
Behavioral: Strength at Home Couples Group — A multiple site randomized trial will compare 10 sessions of PF-RET to 10 sessions of a supportive group therapy. PF-RET focuses on 1) deployment stress and traumatic experiences impacting intimate relationships; 2) communication between intimate partners; 3) conflict and anger management; and 4) closeness and intimacy.
  Other Names: PTSD-Focused Relationship Enhancement Therapy; Returning Veterans and Partners
  Arms: Strength at Home Couples Group
Behavioral: Supportive Group Therapy — A general support group designed to enhance support for healthy relationship building.
  Other Names: Psychological/Behavioral Placebo Control
  Arms: Supportive Group Therapy

SUMMARY:
The purpose of the project is to develop and test a couples-based relationship enhancement group intervention for married or partnered Operation Enduring Freedom (OEF)/Operation Iraqi Freedom (OIF)/Operation New Dawn (OND) veterans to prevent the perpetration of intimate partner aggression (IPA) among participants.

DETAILED DESCRIPTION:
The focus of this project is to produce a well-defined and standardized intervention, labeled Strength at Home Couples Group, that can improve intimate relationship satisfaction, decrease the likelihood of relationship aggression, increase the intimacy and closeness of the relationship, and help with anger management. We hope to learn more about how to improve relationships, how to prevent anger and violence, and about what factors help people successfully complete treatment. Strength at Home Couples Group will incorporate components of several interventions for PTSD and IPA and will target mechanisms implicated in the PTSD-IPA association. The development of this type of integrated intervention is critical due to high rates of PTSD-IPA co-occurrence and the pressing need to efficiently address both problems among military veterans. Specific aims of this project are: (1) to develop and standardize Strength at Home Couples Group for male combat veterans, including the development of a clinician-friendly intervention manual detailing Strength at Home Couples Group, along with intervention adherence measures and therapist training and certification procedures; (2) to test the efficacy of Strength at Home Couples Group for OEF/OIF/OND veterans by conducting a multiple site randomized trial comparing 10 sessions of Strength at Home Couples Group to 10 sessions of a supportive group therapy (ST) condition; and (3) to explore differences in compliance and process factors across conditions.

ELIGIBILITY:
Inclusion Criteria:

* couples must have been in a committed relationship for at least six months
* veterans and their partners must be over the age of 18
* male members of the couple report no occurrence of physical aggression during the last six months in their current relationship on the Revised Conflict Tactics Scale (CTS2; Straus et al, 1996)
* female members of the couple may report that they have engaged in low level aggression during the past six months in their current relationship on the Revised Conflict Tactics Scale (CTS2; Straus et al., 1996)
* one partner of the couple averages at or below a score of 29 on the 6-item Quality of Marriage Index (QMI; Norton, 1983) or a 100 or below on the Dyadic Adjustment Score (DAS; Spanier, 1976), which are cutoff scores often used to distinguish distressed and non-distressed couples (e.g., Slep, Heyman, Williams, Van Dyke, & O'Leary, 2006), or one member of the couple endorses veteran-perpetrated psychological aggression (defined as scoring above the 75%ile on the CTS2 minor psychological aggression subscale, or any endorsement of items on the severe psychological aggression subscale on the CTS2 or the Dominance/Intimidation scale of the Multidimensional Measure of Emotional Abuse, MMEA; Murphy & Hoover, 1999;)
* both members of the couple provide research consent

Exclusion Criteria:

* reading difficulties prevent valid completion of the assessment instruments
* the participant evidences severe organicity or active psychosis
* the participant expresses prominent suicidal or homicidal ideation
* the participant meets diagnostic criteria for alcohol and/or drug dependence, if not in early full remission or sustained partial remission
* female members of the couple report their violence includes the use of weapons during the past six months in their current relationship on the Revised Conflict Tactics Scale (CTS2; Straus et al., 1996)
* violence perpetrated by female members of the couple produces injuries in men
* male members of the couple indicate they are fearful of the female partner
* male members of the couple report they are physically violent in any way during the past six months or severely violent in the past 12 months of their current relationship on the Revised Conflict Tactics Scale (CTS2; Straus et al., 1996)
* male members of the couple have had any bruising or injuries inflicted by the female partner during the past six months in their current relationship. Criteria b through d will be assessed using the Mini-International Neuropsychiatric Interview (MINI; Sheehan et al., 1998) and clinical interview

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 156 (Actual)
Dates: Start 2009-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Evidence of change in incidence and frequency of intimate partner physical assault and psychological aggression assessed by questionnaires and clinical interviews. | Change determined by assessments pre and post treatment, 6 months, 12 months, and 18 months following treatment

SECONDARY OUTCOMES:
Evidence of change in risk factors (i.e. PTSD symptoms, anger, relationship satisfaction) implicated in the development of IPA assessed by questionnaires, clinical interviews, and psychophysiological measurements. | Change determined by assessments pre and post treatment, 6 months, 12 months, and 18 months following treatment

CONTACTS AND LOCATIONS:
Overall Officials: Casey T Taft, Ph.D., Principal Investigator — National Center for PTSD, VA Boston Healthcare System; Suzannah Creech, PhD, Principal Investigator — Providence VA Medical Center
Locations (2):
- United States (2):
  - National Center for PTSD, VA Boston Healthcare System, Boston, Massachusetts
  - Providence VA Medical Center, Providence, Rhode Island

REFERENCES:
- [Background] Norton, R. (1983). Measuring marital quality: A critical look at the dependent variable. Journal of Marriage and the Family, 45, 141-151.
- [Background] Straus, M. A., Hamby, S. L., Boney-McCoy, S., & Sugarman, D. B. (1996). The Revised Conflict Tactics Scales (CTS2): Development and preliminary psychometric data. Journal of Family Issues,17, 283-316.
- [Background] Spanier, G. B. (1976). Measuring dyadic adjustment: New scales for assessing the quality of marriage and similar dyads. Journal of Marriage and the Family, 38, 154-28.
- [Background] Murphy CM, Hoover SA. Measuring emotional abuse in dating relationships as a multifactorial construct. Violence Vict. 1999 Spring;14(1):39-53. PMID 10397625
- [Derived] Taft CT, Creech SK, Gallagher MW, Macdonald A, Murphy CM, Monson CM. Strength at Home Couples program to prevent military partner violence: A randomized controlled trial. J Consult Clin Psychol. 2016 Nov;84(11):935-945. doi: 10.1037/ccp0000129. Epub 2016 Sep 5. PMID 27599224